CLINICAL TRIAL: NCT03344744
Title: Circulating and CSF miRNA Profile in Patients With Acute Aneurysmal Subarachnoid Haemorrhage
Brief Title: miRNA Profile in Aneurysmal Subarachnoid Haemorrhage
Acronym: miRNA
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, George KC Wong, Professor(Clinical), Chinese University of Hong Kong
Other Study IDs: miSAH003
Record Dates: First submitted 2017-10-12; First posted 2017-11-17 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid Haemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SAH with DCI: Aneurysmal subarachnoid haemorrhage patients with delayed cerebral infarction
- SAH nonDCI: Aneurysmal subarachnoid haemorrhage patients without delayed cerebral infarction
- Control: Healthy volunteers

SUMMARY:
The investigators aim to investigate and understand the circulating miRNA profiles after acute aneurysmal subarachnoid haemorrhage and underlying pathological significance.

DETAILED DESCRIPTION:
1. The investigators aim to investigate the miRNA classifier for delayed cerebral infarction after aneurysmal subarachnoid haemorrhage;
2. The investigators aim to investigate the corresponding circulating and CSF miRNA profiles.

ELIGIBILITY:
Inclusion Criteria:

Aneurysmal subarachnoid hemorrhage patients within the first 72 hours or Healthy volunteers

Exclusion Criteria:

Previous neurological diseases such as stroke or dementia

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Acute aneurysmal subarachnoid hemorrhage patients with and without delayed cerebral infarction
  * Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Circulating micro RNA concentrations | Day 3
  Serum micro RNA concentrations

SECONDARY OUTCOMES:
Circulating micro RNA change | Days 1,2,3,7
  Changes of serum micro RNA concentrations between days 1,2,3,7
Cerebrospinal fluid micro RNA concentrations | Day 1,2,3,7
  Cerebrospinal fluid micro RNA concentrations
Cerebrospinal fluid micro RNA change | Days 1,2,3,7
  Changes of cerebrospinal fluid micro RNA concentrations between days 1,2,3,7

CONTACTS AND LOCATIONS:
Overall Officials: George KC Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lu G, Wong MS, Xiong MZQ, Leung CK, Su XW, Zhou JY, Poon WS, Zheng VZY, Chan WY, Wong GKC. Circulating MicroRNAs in Delayed Cerebral Infarction After Aneurysmal Subarachnoid Hemorrhage. J Am Heart Assoc. 2017 Apr 25;6(4):e005363. doi: 10.1161/JAHA.116.005363. PMID 28442458
- [Background] Su XW, Chan AH, Lu G, Lin M, Sze J, Zhou JY, Poon WS, Liu Q, Zheng VZ, Wong GK. Circulating microRNA 132-3p and 324-3p Profiles in Patients after Acute Aneurysmal Subarachnoid Hemorrhage. PLoS One. 2015 Dec 16;10(12):e0144724. doi: 10.1371/journal.pone.0144724. eCollection 2015. PMID 26675167
- [Background] Wong GK, Lam S, Ngai K, Wong A, Mok V, Poon WS; Cognitive Dysfunction after Aneurysmal Subarachnoid Haemorrhage Investigators. Evaluation of cognitive impairment by the Montreal cognitive assessment in patients with aneurysmal subarachnoid haemorrhage: prevalence, risk factors and correlations with 3 month outcomes. J Neurol Neurosurg Psychiatry. 2012 Nov;83(11):1112-7. doi: 10.1136/jnnp-2012-302217. Epub 2012 Jul 31. PMID 22851612